CLINICAL TRIAL: NCT04572711
Title: Prospective Evaluation of Biliary Tissue Sampling with ERCP
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vinay Chandrasekhara, Principal Investigator, Mayo Clinic
Other Study IDs: 20-004079
Record Dates: First submitted 2020-09-09; First posted 2020-10-01 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-11

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Biliary Stricture; Biliary Tract Diseases; Cholangiocarcinoma
MeSH Terms: conditions — Biliary Tract Diseases; Cholangiocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to assess the safety, outcomes and performance characteristics of multiple biliary sampling techniques including but not limited to: single operator cholangioscopy (SOC) directed biopsies, transpapillary biliary biopsies (TPBx), brushings and bile aspiration for cytology and FISH in patients undergoing ERCP.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Diagnosis of indeterminate biliary stricture
* Scheduled clinically indicated ERCP procedure

Exclusion Criteria:

• Adults <18 years, Children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 18 years of age or older who are undergoing ERCP with tissue sampling for an indeterminate biliary stricture will be identified at the time of their scheduled procedure.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Performance characteristics | 1 year after ERCP procedure
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value for the detection of malignancy with each sampling technique
Number of adverse events | Within 30 days of ERCP procedure
  Adverse events after biliary sampling

SECONDARY OUTCOMES:
Healthcare Utilization | through study completion, an average of 2 years
  Number of ERCPs, Radiological studies etc needed before accurate diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials